CLINICAL TRIAL: NCT04876092
Title: A Phase 1b Study of the MALT1 Inhibitor JNJ-67856633 and Ibrutinib in Combination in Relapsed or Refractory B Cell Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: A Study of the MALT1 Inhibitor JNJ-67856633 and Ibrutinib in Combination in B-cell NHL and CLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109010; 67856633LYM1002 (Other: Janssen Research & Development, LLC); 2021-000191-12 (EudraCT Number); 2024-512689-32-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-05-04; First posted 2021-05-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-67856633 and Ibrutinib (Experimental): Participants will receive JNJ-67856633 together with Ibrutinib orally on a 21-day cycle. The dose levels will be escalated based on the dose limiting toxicities (DLT) evaluation by Study Evaluation Team (SET).
  Interventions: Drug: JNJ-67856633; Drug: Ibrutinib

INTERVENTIONS:
Drug: JNJ-67856633 — Participants will receive JNJ-67856633 orally.
Drug: Ibrutinib — Participants will receive Ibrutinib orally.
  Other Names: JNJ-54179060

SUMMARY:
The purpose of this study is to determine the safety and recommended Phase 2 dose (RP2D) of JNJ-67856633 and ibrutinib in combination in participants with B cell non-Hodgkin lymphoma (NHL) and chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
Non-Hodgkin lymphoma (NHL) represents the most frequent hematologic malignancy in the world and represents a diverse set of diseases. JNJ-67856633-ZAF (referred as JNJ-67856633) is an orally bioavailable, potent, and selective first-in-class mucosa-associated lymphoid tissue lymphoma translocation protein-1 (MALT1) inhibitor. JNJ-67856633 binds to an allosteric site on MALT1 with a mixed-type mechanism. Ibrutinib is a first-in-class, orally administered, potent, orally administered covalently binding small-molecule inhibitor of Bruton's tyrosine kinase (BTK), as well as interleukin-2-inducible kinase (ITK), a tyrosine protein (Tec) kinase family member present in T cells. The doses will be escalated in the study and one or more recommended Phase 2 dose (RP2Ds) of JNJ-67856633 will be determined. The study is divided into 3 periods: a screening phase, a treatment phase, and a post-treatment follow-up phase. Efficacy assessments will include radiographic image assessments, positron emission tomography scan, bone marrow assessment, endoscopy etc. Safety assessment like physical examination, vital signs, electrocardiogram (ECG), eastern cooperative oncology group (ECOG) performance status, and adverse events monitoring will be performed during the study. Total duration of the study will be up to 2 years and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Cardiac parameters within the specified range
* Women of childbearing potential must agree to all of the following during the study and for 3 months after the last dose of study drug: a) use a barrier method of contraception; b) use a highly effective contraceptive methods; c) not to donate eggs (ova, oocytes) or freeze them for future use for the purposes of assisted reproduction during the study; d) not to plan to become pregnant; e) not to breast-feed
* Willing and able to adhere to the lifestyle restrictions specified in this protocol
* Participants must have tumor tissue availability
* Adequate organ functions

Exclusion Criteria:

* Known (active) Central Nervous System (CNS) involvement
* Prior treatment with JNJ-67856633 or another MALT1 inhibitor that is associated with disease progression or intolerable toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicity (DLT) | Up to 21 days
  Percentage of Participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematological toxicity or hematological toxicity.
Percentage of Participants with Adverse Events (AEs) by Severity | Up to 2 years and 9 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-67856633 and Ibrutinib | Up to 2 years and 9 months
  Plasma samples will be analyzed to determine concentrations of JNJ-67856633 and Ibrutinib.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- Rigshospitalet, Copenhagen, Denmark
- France (6):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes hotel Dieu, Nantes
  - Hopital St Louis, Paris
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Gustave Roussy, Villejuif
- Poland (2):
  - Pratia MCM Krakow, Krakow
  - Centrum Medyczne Pratia Poznan, Skorzewo
- Universitetssjukhuset Lund, Onkologiska Kliniken, Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency